CLINICAL TRIAL: NCT02588404
Title: The Predictive Value of TMPRSS2-ERG Fusion in High Risk Prostate Cancer Patient with Biochemical Failure Status Post Salvage or Radical Radiation Therapy (PCS VIII)
Brief Title: The Predictive Value of TMPRSS2-ERG Fusion in High Risk Prostate Cancer Patient
Status: Withdrawn | Type: Observational
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Tamim Niazi, Principal investigator, Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: Fusion study
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — luprolide acetate gel depot; Leuprolide; Triptorelin Pamoate; Goserelin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Areas of prostate tumor will be identified by the pathologist of the study. This will then be excised from the paraffin block using a tissue microarray punch. Two punches will be acquired: one for RNA extraction and one for DNA extraction. RNA and DNA will be extracted using the RecoverAll Nucleic Acid Isolation Kit (Ambion). Standard protocol for the isolation of nucleic acids will be used differing only in the time of protease digestion such that RNA is isolated after a short incubation (30 minutes), while DNA is isolated after a longer incubation (overnight).
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Drug: LHRH therapy — These patients will be treated with LHRH agonist as standard therapy.
  Other Names: Eligard, Lupron, Trelstar, and Zoladex

SUMMARY:
The objective of this study is to evaluate the predictive value of TMPRSS2-ERG gene fusion in patients with prostate cancer treated with radiation and hormonal therapy.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the predictive value of TMPRSS2-ERG gene fusion in prostate patients who have been treated with hormonal and radiation treatment after biochemical failure

Original biopsy slides of 65 patients will be collected and reviewed. A tissue used to test and map DNA fragments will be constructed from patients who underwent radiation therapy. RNA and DNA will be extracted from each slide. This study, if positive, will establish the predictive value of TMPRSS2-ERG gene fusion in prostate cancer patients. It can lead to believe that high-risk prostate cancer patients will benefit from a more aggressive treatment.

An endpoint of this study is to evaluate the relation between the Gleason score and the TMPRSS2-ERG gene fusion. Another is to evaluate the relation between the T-stage and TMPRSS2-ERG gene fusion.

ELIGIBILITY:
Inclusion Criteria: One of the following

* T3a +
* PSA > 20
* Gleason 8 or higher
* Karnofsky performance status ≥ 70.
* Signed study-specific informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The original slides of 65 patients with informed consent will be reviewed. Assuming 50% Gene-fusion carrier rate, patients with and without markers under the investigation will be accrued into this study. The investigators at the treating institutions will submit paraffin-embedded tissue blocks from the original pre-treatment diagnostic prostatic biopsy, which will be reviewed to confirm the Gleason score and to record other histopathologic features, such as the extent of tumor in the biopsies, the number of positive biopsies, and mitotic index. The block must be clearly labeled with the protocol and case number. A tissue microarray (TMA) containing cores representing clinically localized prostate cancers will be constructed from 60 men who underwent radical radiation therapy. Three cores (0.6mm in diameter) will be taken from each representative tissue block to construct the TMA. Detailed clinical, pathological, and TMA data will be maintained on a secure database.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with biochemical failure showing presence of TMPRSS2-ERG gene fusion. | recruitment over 4 years
  Biopsy samples of patients treated for high risk prostate cancer with radical radiation and hormonal therapy (LHRH) will be tested to evaluate the predictive value of the TMPRSS2-ERG gene fusionThe results between the two groups will be compared to see if either DNA changes are an indicator of LHRH refractoriness